CLINICAL TRIAL: NCT06813846
Title: Assessment of Pink Esthetic Score After Using Two Papilla Reconstruction Exposure Techniques Versus Mid-Crestal Sulcular Incision in Second Stage Implant Surgery: a Randomized Controlled Clinical Trail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sarah Rajab, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-035
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Papilla Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- "I" shaped incision (Experimental): A Labial horizontal incision with a #15c blade will be performed mesiodistally 0.5-1.0 mm inside from the labial border of the implant. A horizontal incision will also be performed, parallel to the buccal side, on the palatal side, which is in contact with the palatal border line of the implant different from the labial side. Another incision will be done bucco-lingually over the implant midline perpendicular to the horizontal incision lines performed on the labial and palatal sides. The flap will be reflected with care and the implant will be exposed to remove the cover screw. The healing abutment will be connected and both flaps will be folded up alongside the healing abutment intending them to heal without suture.
  Interventions: Procedure: "I" shaped incision
- Split-Finger Procedure (Experimental): The surgical technique first designs 3 interlacing "fingers" over and adjacent to each implant site and will be extended around each adjacent tooth. · A sulcular incision will be made 2 to 3 mm to the palatal side from each tooth with a loop design (at least 2.0-2.5 mm) adjacent to the implant location. · The incisions will then be joined facially with a semicircular incision at the preplanned free tissue margin of the implant crown. · The facial "fingers" will be elevated to the desired interimplant height for the papillae. The middle "palatal finger" will then be split and reflected to the respective mesial and distal sides (each is at least 2.0-2.5 mm wide). · The soft tissue maintains its elevated position with a permucosal extension or a final prosthetic abutment that is extended through the soft tissue. · A modified vertical mattress suture will then be used to suture each papilla using 4-0 or 5-0 Gut or Vicryl sutures.
  Interventions: Procedure: Split-Finger Procedure
- Mid-Crestal Sulcular Incision (Active Comparator): A long incision over the crest and midway between buccolingual aspect through the gingiva from the site of the distal implant in mesial direction with intra-sulcular incisions in the teeth adjected to the implant site · Following a full or partial thickness flap is raised to establish access to cover screw.
  Interventions: Procedure: Mid-Crestal Sulcular Incision

INTERVENTIONS:
Procedure: Mid-Crestal Sulcular Incision — A long incision over the crest and midway between buccolingual aspect through the gingiva from the site of the distal implant in mesial direction with intra-sulcular incisions in the teeth adjected to the implant site · Following a full or partial thickness flap is raised to establish access to cover screw.
  Arms: Mid-Crestal Sulcular Incision
Procedure: Split-Finger Procedure — The surgical technique first designs 3 interlacing "fingers" over and adjacent to each implant site and will be extended around each adjacent tooth. · A sulcular incision will be made 2 to 3 mm to the palatal side from each tooth with a loop design (at least 2.0-2.5 mm) adjacent to the implant location. · The incisions will then be joined facially with a semicircular incision at the preplanned free tissue margin of the implant crown. · The facial "fingers" will be elevated to the desired interimplant height for the papillae. The middle "palatal finger" will then be split and reflected to the respective mesial and distal sides (each is at least 2.0-2.5 mm wide). · The soft tissue maintains its elevated position with a permucosal extension or a final prosthetic abutment that is extended through the soft tissue. · A modified vertical mattress suture will then be used to suture each papilla using 4-0 or 5-0 Gut or Vicryl sutures.
  Arms: Split-Finger Procedure
Procedure: "I" shaped incision — A Labial horizontal incision with a #15c blade will be performed mesiodistally 0.5-1.0 mm inside from the labial border of the implant. A horizontal incision will also be performed, parallel to the buccal side, on the palatal side, which is in contact with the palatal border line of the implant different from the labial side. Another incision will be done bucco-lingually over the implant midline perpendicular to the horizontal incision lines performed on the labial and palatal sides. The flap will be reflected with care and the implant will be exposed to remove the cover screw. The healing abutment will be connected and both flaps will be folded up alongside the healing abutment intending them to heal without suture.
  Arms: "I" shaped incision

SUMMARY:
The purpose of this randomized clinical trial is to assess the pink esthetic score with three different techniques in second-stage implant surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who already received implants in the anterior and premolar region
2. All implants were placed 4 months prior to uncovering in the mandible and 6 months prior to uncovering in the maxilla.
3. Patients with good oral hygiene
4. Medically free patients
5. Adequate keratinized tissue

Exclusion Criteria:

1. Acute infection
2. Occlusal trauma
3. Smokers
4. Pregnancy and lactation
5. Severe gag reflex

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | 6 Months
  Pink esthetic score will be recorded for five variables: "mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue color and texture at the facial aspect of the implant site". A score of 2, 1, or 0 will be assigned to all five PES parameters. The two papillary scores (mesial and distal) will be assessed for the complete presence (score 2), incomplete presence (score 1) or absence (score0) of papillary tissue. The curvature of the facial soft tissue line, also defined as the line of emergence of the implant restoration from the soft tissues, will be evaluated as being identical (score 2 ), slightly different (score 1), or markedly different (score 0) compared to the natural control tooth and thus, provided a natural
  symmetrical or disharmonious appearance and in comparison to the contralateral tooth in terms of an identical vertical level (score 2), a slight (<1 mm) discrepancy (score 1), or a major (>1 mm) discrepancy

SECONDARY OUTCOMES:
Healing Index | 1 Month
  The healing index included five clinical outcome parameters: tissue color (percent of red vs pink gingiva), presence of bleeding on palpation, presence of granulation tissue, incision margin (epithelization and connective tissue exposure), and presence of suppuration. The final score ranged from 0 (poor healing) to 5 (excellent healing).
Volumetric Changes | baseline, 3, 6 and 9 months
  To assess the volumetric differences between the baseline, 3, 6 and 9 months postoperatively. Digital replicas will be produced resembling various time intervals during treatment. Superimposing the different replicas of each case utilizing the best fit algorithm by using reference points from the tooth surfaces. The implant site region will be delineated by the mucogingival line, the mesial and distal papillary midline and the alveolar crest. Thus, alterations in volume between the digitized superimposed replicas could be recorded.
Visual analogue scale | 2 Weeks
  Pain score is reported by the patient directly through The Visual Analogue Scale score (from 0 to 10. 0: no pain, 1: minimal pain, 5: moderate pain, 10: severe pain)
The Oral health impact profile (OHIP-14 questionnaire) | 6 Months
  Will be used to assess limitation of function, pain, discomfort, social, psychological, physical disability, and general satisfaction. The OHIP-14 utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often). A lower score in any of the five categories indicates higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - The British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided